CLINICAL TRIAL: NCT06514950
Title: Yoga Breath Training to Improve Cardiorespiratory Synchrony in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, PhD, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024P001385
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
Keywords: SCI, Ujjayi, yogic breathing, pranayama
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This study is a small (N = 20) prospective cohort with a single unblinded intervention of Ujjayi resistance breathing at Spaulding Hospital Cambridge. Participants will have two lab visits: a baseline assessment and a post-intervention assessment six weeks later, each lasting about 4 hours. Cardiovascular and respiratory variables will be recorded during controlled and uncontrolled breathing. Coaching sessions in weeks 1 and 4 and virtual sessions via Zoom will train participants in the intervention, focusing on resistance breathing techniques. Participants will practice these techniques twice daily at home (~20 min/day) over six weeks, totaling ~10 hours of in-person lab time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ujjayi yogic breathing training (Experimental): This study will be a small (N = 20) prospective cohort study with a single unblinded intervention of Ujjayi resistance breathing.
  Interventions: Behavioral: Ujjayi Yogic Breathing

INTERVENTIONS:
Behavioral: Ujjayi Yogic Breathing — Participants will undergo 6 weeks of resistive yogic breathing (Ujjayi) upon exhalation (first three weeks) and upon inhalation and exhalation (second three weeks).
  Other Names: resistive breathing

SUMMARY:
The goal of this interventional study is to understand how regular yogic breathing practice, particularly a slow resistive yogic breathing technique called Ujjayi, would benefit individuals between the ages of 18 and 60 with spinal cord injuries. Previously yogic breathing has shown to improve respiratory function and sleep- we'd like to explore this further.

The main questions this study aims to answer are:

* How does Ujjayi breathing affect breathing patterns in individuals with spinal cord injuries?
* How does Ujjayi breathing affect lung function in individuals with spinal cord injuries?
* How does Ujjayi breathing affect the part of the nervous system responsible for ventilatory control in individuals with spinal cord injuries?
* How does Ujjayi breathing affect ventilatory perfusion (how well air and blood flow match in the lungs for efficient gas exchange) in individuals with spinal cord injuries?
* How does Ujjayi breathing affect sleep quality in individuals with spinal cord injuries?

Participants will undergo six weeks of training in Ujjayi breathing. Before and after this period, they will visit the lab for measurements of blood pressure, pulse, blood oxygen levels, and breathing. They will also perform several tests:

* Pulmonary function testing to assess lung capacity and respiratory muscle strength.
* Pace breathing frequency to four pre-recorded audio files at various breathing rates.
* Breathing exercises involving higher levels of carbon dioxide for a short time.
* Breathing exercises involving lower levels of oxygen for a short time.
* At-home sleep evaluation.

Between the two laboratory testing sessions, participants will practice yogic resistance breathing (Ujjayi breathing) for six weeks.

DETAILED DESCRIPTION:
This study investigates the impact of a type of slow-resistive yogic breathing, Ujjayi Pranayama, on cardiopulmonary function in 20 men and women aged 18-60 with spinal cord injuries classified under the American Spinal Injury Association Impairment Scale (AIS) score of A, B, or C. Participants will undergo baseline and post-intervention laboratory assessments over six weeks at Spaulding Hospital Cambridge, with cardiovascular and respiratory measurements taken during controlled and uncontrolled breathing conditions. Ujjayi Pranayama training, focusing on resistance breathing during exhalation and inhalation, will include coaching sessions in weeks 1 and 4, supplemented by virtual support for home practice (~20 min, twice daily). The study aims to determine whether regular yogic breathing practice enhances sleep quality, hypercapnic ventilatory response, and overall cardiopulmonary synchrony, potentially reducing respiratory and cardiovascular risks associated with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* American Spinal Injury Association Impairment Scale (AIS) score of A, B, or C
* Aged 18-60 years
* Wheelchair user
* Medically stable and able to follow directions
* Body mass index of 18.5 - 35 kg/m2

Exclusion Criteria:

* Resting blood pressure of >140/90 mmHg
* Current use of tobacco or cardioactive medications (except medication to support blood pressure)
* Significant arrhythmia
* Bleeding disorder
* Pulmonary disease
* Coronary artery disease
* Diabetes
* Renal disease
* Cancer
* Epilepsy or other neurological diseases
* Current use of CPAP/BIPAP
* Has smartphone or device incompatible with the PranaTM application

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Ventilatory pattern after regular Ujjayi breathing | Change in ventilatory pattern, Time Frame: Baseline, Week 6
  Ventilatory patterns measured as rate and regularity by breathing belts (pneumobelts). A normal respiratory rate for an adult at rest is 12 to 18 breaths per minute.
Pulmonary function after regular Ujjayi breathing | Change in pulmonary function, Time Frame: Baseline, Week 6
  Pulmonary function measured by spirometry, maximal voluntary ventilation, and maximum inspiratory and expiratory pressures. Results will be reported as forced vital capacity (FVC), Forced Expiratory Volume in 1 second (FEV1), FEV1/FVC ratio, Peak Expiratory Flow (PEF), and Forced Expiratory Flow (FEF) 25%-75%. An absolute range cannot be provided as it depends on various factors such as injury level, completeness of injury, age, race, and sex. In healthy adults, MVV is typically around 120-170 liters per minute (L/min).
Central and peripheral chemosensitivity after regular Ujjayi breathing | Change in central and peripheral chemosensitivity, Time Frame: Baseline, Week 6
  The Read rebreathing method assesses neural drive to breathe and CO2 sensitivity (central chemosensitivity). A three-way valve connects the breathing circuit to room air or 95% O2-5% CO2. Subjects exhale to functional residual capacity, then rebreathe until PETCO2 reaches 55 mmHg, they can't continue, SPO2 drops below 95%, or 10 minutes elapse. Peripheral chemosensitivity uses brief exposures to hypercapnic (10% CO2, 21% O2) or hypoxic gas (pure nitrogen). Ventilatory response is measured over up to 30 seconds, followed by room air. Each test takes about 15 minutes. Tests are conducted seated and supine. Chemosensitivity is measured by plotting ventilation against pulmonary gas levels.
Ventilatory perfusion after regular Ujjayi breathing | Change in ventilatory perfusion, Time Frame: Baseline, Week 6
  Ventilatory perfusion will be calculated from mixed expired and end tidal CO2 measures. The V/Q ratio in healthy lungs is close to 1- this means that ventilation (V) matches perfusion (Q) almost perfectly in well-ventilated alveoli. Certain pathologies could increase or decrease the V/Q ratio.
Sleep quality after regular Ujjayi breathing | Change in sleep quality, Time Frame: Baseline, Week 6
  Sleep quality is assessed using two methods: the PROMIS Sleep Disturbance Short Form and NoxA1 polysomnography. The PROMIS survey provides raw scores that are converted into T-scores. T-scores falling between 40 and 59 indicate average sleep disturbance levels, considered within the normal range. Scores above 60 suggest more sleep disturbances than average, while scores below 39 indicate less disturbance compared to average.
  NoxA1 polysomnography records several parameters including EEG waves for sleep stages, wake after onset, nocturnal disturbances, maximum and minimum heart rates at rest, breathing rates, limb movements, teeth grinding (monitored via chin movement sensors), blood oxygen saturation, and respiratory patterns.

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, MS, PhD, Principal Investigator — Harvard Medical School/Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shields RK. Muscular, skeletal, and neural adaptations following spinal cord injury. J Orthop Sports Phys Ther. 2002 Feb;32(2):65-74. doi: 10.2519/jospt.2002.32.2.65. PMID 11838582
- [Background] Zimmer MB, Nantwi K, Goshgarian HG. Effect of spinal cord injury on the respiratory system: basic research and current clinical treatment options. J Spinal Cord Med. 2007;30(4):319-30. doi: 10.1080/10790268.2007.11753947. PMID 17853653
- [Background] Tollefsen E, Fondenes O. Respiratory complications associated with spinal cord injury. Tidsskr Nor Laegeforen. 2012 May 15;132(9):1111-4. doi: 10.4045/tidsskr.10.0922. English, Norwegian. PMID 22614314
- [Background] Burns SP, Kapur V, Yin KS, Buhrer R. Factors associated with sleep apnea in men with spinal cord injury: a population-based case-control study. Spinal Cord. 2001 Jan;39(1):15-22. doi: 10.1038/sj.sc.3101103. PMID 11224009
- [Background] van den Berg ME, Castellote JM, de Pedro-Cuesta J, Mahillo-Fernandez I. Survival after spinal cord injury: a systematic review. J Neurotrauma. 2010 Aug;27(8):1517-28. doi: 10.1089/neu.2009.1138. PMID 20486810
- [Background] Waddimba AC, Jain NB, Stolzmann K, Gagnon DR, Burgess JF Jr, Kazis LE, Garshick E. Predictors of cardiopulmonary hospitalization in chronic spinal cord injury. Arch Phys Med Rehabil. 2009 Feb;90(2):193-200. doi: 10.1016/j.apmr.2008.07.026. PMID 19236973
- [Background] Tran K, Hukins C, Geraghty T, Eckert B, Fraser L. Sleep-disordered breathing in spinal cord-injured patients: a short-term longitudinal study. Respirology. 2010 Feb;15(2):272-6. doi: 10.1111/j.1440-1843.2009.01669.x. Epub 2009 Nov 30. PMID 19947995
- [Background] Burns SP, Rad MY, Bryant S, Kapur V. Long-term treatment of sleep apnea in persons with spinal cord injury. Am J Phys Med Rehabil. 2005 Aug;84(8):620-6. doi: 10.1097/01.phm.0000171008.69453.b9. PMID 16034232
- [Background] Raguindin PF, Frankl G, Itodo OA, Bertolo A, Zeh RM, Capossela S, Minder B, Stoyanov J, Stucki G, Franco OH, Muka T, Glisic M. The neurological level of spinal cord injury and cardiovascular risk factors: a systematic review and meta-analysis. Spinal Cord. 2021 Nov;59(11):1135-1145. doi: 10.1038/s41393-021-00678-6. Epub 2021 Aug 20. PMID 34417550
- [Background] Schuster AK, Fischer JE, Thayer JF, Mauss D, Jarczok MN. Decreased heart rate variability correlates to increased cardiovascular risk. Int J Cardiol. 2016 Jan 15;203:728-30. doi: 10.1016/j.ijcard.2015.11.027. Epub 2015 Nov 6. No abstract available. PMID 26587729
- [Background] Solinsky R, Vivodtzev I, Hamner JW, Taylor JA. The effect of heart rate variability on blood pressure is augmented in spinal cord injury and is unaltered by exercise training. Clin Auton Res. 2021 Apr;31(2):293-301. doi: 10.1007/s10286-020-00677-2. Epub 2020 Mar 12. PMID 32166421
- [Background] Ely MR, Schleifer GD, Singh TK, Baggish AL, Taylor JA. Exercise Training Does Not Attenuate Cardiac Atrophy or Loss of Function in Individuals With Acute Spinal Cord Injury: A Pilot Study. Arch Phys Med Rehabil. 2023 Jun;104(6):909-917. doi: 10.1016/j.apmr.2022.12.001. Epub 2022 Dec 23. PMID 36572202
- [Background] Solinsky R, Mercier H, Picard G, Taylor JA. Cardiometabolic Effects of High-Intensity Hybrid Functional Electrical Stimulation Exercise after Spinal Cord Injury. PM R. 2021 Sep;13(9):937-944. doi: 10.1002/pmrj.12507. Epub 2020 Dec 4. PMID 33027550
- [Background] Chou RC, Taylor JA, Solinsky R. Effects of hybrid-functional electrical stimulation (FES) rowing whole-body exercise on neurologic improvement in subacute spinal cord injury: secondary outcomes analysis of a randomized controlled trial. Spinal Cord. 2020 Aug;58(8):914-920. doi: 10.1038/s41393-020-0445-3. Epub 2020 Feb 24. PMID 32094516
- [Background] Bertisch SM, Hamner J, Taylor JA. Slow Yogic Breathing and Long-Term Cardiac Autonomic Adaptations: A Pilot Study. J Altern Complement Med. 2017 Sep;23(9):722-729. doi: 10.1089/acm.2016.0074. Epub 2017 Apr 18. PMID 28418684
- [Background] Chiodo AE, Sitrin RG, Bauman KA. Sleep disordered breathing in spinal cord injury: A systematic review. J Spinal Cord Med. 2016 Jul;39(4):374-82. doi: 10.1080/10790268.2015.1126449. Epub 2016 Mar 15. PMID 27077573
- [Background] Aboussouan LS. Sleep-disordered Breathing in Neuromuscular Disease. Am J Respir Crit Care Med. 2015 May 1;191(9):979-89. doi: 10.1164/rccm.201412-2224CI. PMID 25723731
- [Background] Norrbrink Budh C, Hultling C, Lundeberg T. Quality of sleep in individuals with spinal cord injury: a comparison between patients with and without pain. Spinal Cord. 2005 Feb;43(2):85-95. doi: 10.1038/sj.sc.3101680. PMID 15570322
- [Background] Somers VK, White DP, Amin R, Abraham WT, Costa F, Culebras A, Daniels S, Floras JS, Hunt CE, Olson LJ, Pickering TG, Russell R, Woo M, Young T; American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology; American Heart Association Stroke Council; American Heart Association Council on Cardiovascular Nursing; American College of Cardiology Foundation. Sleep apnea and cardiovascular disease: an American Heart Association/american College Of Cardiology Foundation Scientific Statement from the American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology, Stroke Council, and Council On Cardiovascular Nursing. In collaboration with the National Heart, Lung, and Blood Institute National Center on Sleep Disorders Research (National Institutes of Health). Circulation. 2008 Sep 2;118(10):1080-111. doi: 10.1161/CIRCULATIONAHA.107.189375. Epub 2008 Aug 25. No abstract available. PMID 18725495
- [Background] Sankari A, Vaughan S, Bascom A, Martin JL, Badr MS. Sleep-Disordered Breathing and Spinal Cord Injury: A State-of-the-Art Review. Chest. 2019 Feb;155(2):438-445. doi: 10.1016/j.chest.2018.10.002. Epub 2018 Oct 12. PMID 30321507
- [Background] Burns SP, Little JW, Hussey JD, Lyman P, Lakshminarayanan S. Sleep apnea syndrome in chronic spinal cord injury: associated factors and treatment. Arch Phys Med Rehabil. 2000 Oct;81(10):1334-9. doi: 10.1053/apmr.2000.9398. PMID 11030498
- [Background] Leduc BE, Dagher JH, Mayer P, Bellemare F, Lepage Y. Estimated prevalence of obstructive sleep apnea-hypopnea syndrome after cervical cord injury. Arch Phys Med Rehabil. 2007 Mar;88(3):333-7. doi: 10.1016/j.apmr.2006.12.025. PMID 17321826
- [Background] Bascom AT, Sankari A, Badr MS. Spinal cord injury is associated with enhanced peripheral chemoreflex sensitivity. Physiol Rep. 2016 Sep;4(17):e12948. doi: 10.14814/phy2.12948. PMID 27597767
- [Background] Raurich JM, Rialp G, Llompart-Pou JA, Ayestaran I, Perez-Barcena J, Ibanez J. Respiratory CO(2) response in acute cervical spinal cord injury (CO(2) response in spinal cord injury). Spinal Cord. 2014 Jan;52(1):39-43. doi: 10.1038/sc.2013.115. Epub 2013 Oct 8. PMID 24100664
- [Background] Stanescu DC, Nemery B, Veriter C, Marechal C. Pattern of breathing and ventilatory response to CO2 in subjects practicing hatha-yoga. J Appl Physiol Respir Environ Exerc Physiol. 1981 Dec;51(6):1625-9. doi: 10.1152/jappl.1981.51.6.1625. PMID 6798002